CLINICAL TRIAL: NCT06375187
Title: A Phase I Study to Evaluate the Safety and Efficacy of Engineering Tumor Infiltrating Lymphocytes Injection (GC203 TIL)in Patients With Advanced Malignant Solid Tumors
Brief Title: A Study of GC203 TIL in Advanced Malignant Solid Tumors
Acronym: KUNLUN-001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Juncell Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC203 TIL-ST-Ⅰ
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor; Gynecologic Cancer; Breast Cancer; Gastrointestinal Cancer; Lung Cancer
Keywords: Adoptive cell therapy; Tumor Infiltrating Lymphocytes
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Engineering Tumor Infiltrating Lymphocytes Injection (GC203 TIL)
  Interventions: Biological: Engineering Tumor Infiltrating Lymphocytes

INTERVENTIONS:
Biological: Engineering Tumor Infiltrating Lymphocytes — A tumor sample is resected from each participant and cultured ex vivo to generate the engineered tumor infiltrating lymphocytes. After lymphodepletion, patients are infused GC203 TIL followed low-dose PD-1 antibody.
  Other Names: GC203 TIL

SUMMARY:
A clinical trial to assess the safety and efficacy of engineered Tumor Infiltrating Lymphocytes (TIL) for the treatment of Advanced Malignant Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* 1. In the opinion of the Investigator, patients must be able to sign the ICF and complete all study-required procedures.

  2. Patients must be ≥18 and ≤75 years of age at the time of consent. 3. Patients with advanced metastatic solid tumors with clear pathological diagnosis have failed standard therapy (standard therapy is defined as existing guidelines and consensus recommended therapy [including but not limited to chemotherapeutic therapy, radiotherapy, mutation-targeted therapy, immunotherapy, and surgery]) , including but not limited to gynecological tumors (ovarian cancer, endometrial cancer, cervical cancer), breast cancer, gastrointestinal Cancer, lung cancer.

  4. Patients have feasible tissue areas for tumor resection/puncture to generate GC203 TIL, the total volume of the tissue > 400mm3, and the lesion has not received local treatment (such as radiotherapy, radiofrequency therapy, oncolytic virus, etc.) or has progressed after local treatment; 5. At least one measurable target lesion before preconditioning, as defined by RECIST1.1.

  6. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

  7. Patients must have an estimated life expectancy of ≥3 months. 8. Patients must have the following hematologic parameters, Coagulation functions and hepatic and renal function:
  * Absolute Neutrophil Count (ANC)≥1.0×10^9/L;
  * Absolute Lymphocyte Count(ALC)≥0.5×10^9/L;
  * Platelet≥80×10^9/L；
  * International Normalized Ratio（INR）≤1.5×ULN;
  * Activated Partial Thromboplastin Time（APTT）≤1.5×ULN;
  * Serum Creatinine (Scr)≤1.5mg/dL (or 132.6μmol/L) or Creatinine Clearance≥60mL/min
  * Urinalysis: urine protein less than 2+, or 24-hour urine protein <1g;
  * Alanine aminotransferase(AST/SGOT) ≤3×ULN;
  * Alanine aminotransferase (ALT/SGPT) ≤3×ULN;
  * Total Bilirubin(TBIL)≤1.5×ULN； 9. Women of child-bearing potential (WCBP), must have a negative serum pregnancy test prior to treatment. All sexually active WCBP and all sexually active male subjects must agree to use effective methods of birth control throughout the study.

    10. Patients must have no contraindications for surgery or biopsy. 11. Patients have good compliance and be able to adhere to research access plans and other protocol requirements.

Exclusion Criteria:

1. Participate in clinical trials of other drugs or biologic therapies within 4 weeks before enrollment;
2. Participants who have had a history of allogeneic T cell therapy; gene engineering autologous cell therapy within 1 years.
3. Patients who have received systemic antitumor therapy within 4 weeks.
4. Patients who have had another primary malignancy within the previous 5 years
5. Patients who have received a live or attenuated vaccination within 28 days prior to the start of treatment
6. Patients with a history of hypersensitivity to any component of the study drugs
7. Patients who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Maximal Tolerance Dose | Up to Day 28
Dose Limiting Toxicity | Up to Day 28
Adverse Events | Maximum 360 days

SECONDARY OUTCOMES:
Objective Response Rate | Every 6 weeks for 12 months
  Evaluate the efficacy endpoints of ORR by the investigator with RECIST v1.1 and iRECIST
Duration of Response | Every 6 weeks for 12 months
  Evaluate the efficacy endpoints of DoR by the investigator with RECIST v1.1 and iRECIST
Disease Control Rate | Every 6 weeks for 12 months
  Evaluate the efficacy endpoints of DCR by the investigator with RECIST v1.1 and iRECIST
Progression-Free Survival | Every 6 weeks for 12 months
  Evaluate the efficacy endpoints of PFS by the investigator with RECIST v1.1 and iRECIST
Overall Survival | Every 6 weeks for 12 months
  Evaluate the efficacy endpoints of OS by the investigator with RECIST v1.1 and iRECIST
Quality of Life Assessment | Every 6 weeks for 12 months
  Evaluate with EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No